CLINICAL TRIAL: NCT03322293
Title: Tolerability and Efficacy of Daylight Aminolevulinic-acid-photodynamic Therapy (ALA-PDT) Compared With Conventional ALA-PDT for Treatment of Actinic Keratosis on the Face or Scalp
Brief Title: Daylight Photodynamic Therapy for Actinic Keratosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Daylight PDT
Record Dates: First submitted 2017-05-09; First posted 2017-10-26 (Actual); Results first posted 2019-10-04 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses; photodynamic therapy; aminolevulinic acid; precancerous skin lesion
MeSH Terms: conditions — Keratosis, Actinic | interventions — Aminolevulinic Acid; Solutions

STUDY DESIGN:
Intervention Model Description: Randomized (1:1:1), single-blind controlled trial with parallel group design
Who Masked: Investigator
Masking Description: This is a single-blinded study, as the subject cannot be blinded to treatment. Disease assessments and aminolevulinic acid (ALA) application will be performed by the blinded investigator. History, concomitant medications, randomization, light exposure, symptom assessment, and Skindex-16 will be administered by the unblinded study coordinator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- A. Conventional arm (Active Comparator): This is considered the standard of care arm for photodynamic therapy for the treatment of actinic keratosis. This treatment arm includes: Acetone preparation, ALA topical application, 1 hour incubation, 16 minutes 40 seconds (16:40) BLU-U exposure, application of sunscreen.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: BLU-U blue light phototherapy illuminator
  Interventions: Drug: Aminolevulinic Acid Topical 20% Topical Solution; Device: BLU-U blue light phototherapy illuminator
- B. Combination arm (Experimental): This treatment arm combines standard of care BLU-U exposure and daylight exposure. This treatment arm includes: Acetone preparation, ALA topical application, 15 minute incubation, 16:40 BLU-U exposure, application of sunscreen, 45 minute daylight exposure.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: BLU-U blue light phototherapy illuminator
  Interventions: Drug: Aminolevulinic Acid Topical 20% Topical Solution; Device: BLU-U blue light phototherapy illuminator
- C. Daylight arm (Experimental): This is the experimental arm. This treatment arm includes: Acetone preparation, ALA topical application, 15 minute incubation, application of sunscreen, 1 hour daylight exposure.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: none
  Interventions: Drug: Aminolevulinic Acid Topical 20% Topical Solution

INTERVENTIONS:
Drug: Aminolevulinic Acid Topical 20% Topical Solution — PDT involves the topical application of aminolevulinic acid (ALA), or one of its derivatives, as a photosensitizing agent. Subjects will receive ALA in all treatment arms (A, B, and C).
Device: BLU-U blue light phototherapy illuminator — Depending on the treatment arm, subjects will either receive BLU-U exposure or not. Treatment arms A and B have BLU-U exposure and treatment arm C does not.
  Arms: A. Conventional arm; B. Combination arm

SUMMARY:
This is a randomized, single-blind controlled trial with parallel group design to determine whether daylight photodynamic therapy (PDT) affords a reduction in treatment symptoms of pain, burning, and pruritus as measured by 1) symptom level during the treatment period and 2) pain at the end of treatment exposure.

DETAILED DESCRIPTION:
Actinic keratoses (AK) are common precancerous skin lesions that arise on sun-damaged skin. Treatment is aimed at preventing progression to cutaneous squamous cell carcinoma (SCC). First-line therapy for clinically apparent lesions includes cryotherapy and curettage; and field therapy options are topical 5-fluorouracil, imiquimod, ingenol mebutate, and photodynamic therapy (PDT). PDT involves the topical application of aminolevulinic acid (ALA), or one of its derivatives, as a photosensitizing agent. In response, rapidly proliferating, dysplastic cells preferentially accumulate protoporphyrin IX (PpIX). When PpIX is activated by blue or red light, singlet oxygen species are produced, resulting in cell death. PDT is beneficial due to its brief treatment course and efficacy in clearing AK. However, its main drawbacks are the adverse effects of pain, burning, pruritus, erythema, crusting, and inflammation associated with treatment. While conventional PDT uses red or blue artificial light to activate a high concentration of accumulated protoporphyrins, daylight PDT uses natural daylight to activate lower levels of protoporphyrins in a continuous manner. Daylight PDT, when compared with conventional PDT, has been associated with significantly less pain while achieving comparable efficacy for the treatment of AK. Daylight PDT is also more cost-effective and reduces the amount of time spent in clinic. Previous randomized studies comparing daylight PDT with conventional PDT have largely used methyl-aminolevulinate as the photosensitizer, have been intra-individual comparative studies, and have been performed in Nordic countries. Because the effective light dose from natural daylight depends on geographic location and seasonal and weather changes, randomized trials in different geographic and environmental conditions are of interest. The proposed randomized clinical trial investigates the tolerability and efficacy of daylight ALA-PDT for the treatment of AK in San Francisco for the first time; subjects will be randomized to various treatment arms, as opposed to previous split-face and intra-individual studies.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years old.
* Subjects must be able to read, sign, and understand the informed consent
* Subjects have at least 4 and no more than 20 clinically typical, visible actinic keratoses in the target treatment area on the face or scalp.
* Subject must be willing to forego any other treatments for AK in the treatment area on the face or scalp, during the study period, and for 14 days prior to screening; including cryotherapy, topical 5-fluorouracil, imiquimod, and ingenol mebutate.
* Subjects who have previously received PDT must undergo at least an 8-week washout period prior to enrollment in study.
* Subject must be willing and able to participate in the study and to comply with all study requirements including concomitant medication and other treatment restrictions, and telephone interview.
* If subject is a female of childbearing potential she must have a negative urine pregnancy test result prior to study treatment initiation and must agree to use an approved method of birth control while enrolled in the study. Women who are pregnant, lactating, or planning to become pregnant during the study period are excluded from the study.

Exclusion Criteria:

* Subjects with any dermatologic disease in the treatment area that may be exacerbated by the treatment proposed or that might impair the evaluation of AKs.
* Subjects who are currently participating in another clinical study or have completed another clinical study with an investigational drug or device on the study area within 30 days prior to study treatment initiation.
* Subjects with any medical condition that, in the opinion of the investigator, makes the patient unsuitable for the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Arron, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Dermatology, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- A. Conventional Arm: This is considered the standard of care arm for photodynamic therapy for the treatment of actinic keratosis. This treatment arm includes: Acetone preparation, ALA topical application, 1 hour incubation, 16 minutes 40 seconds (16:40) BLU-U exposure, application of sunscreen.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: BLU-U blue light phototherapy illuminator
  Aminolevulinic Acid Topical 20% Topical Solution: PDT involves the topical application of aminolevulinic acid (ALA), or one of its derivatives, as a photosensitizing agent. Subjects will receive ALA in all treatment arms (A, B, and C).
  BLU-U blue light phototherapy illuminator: Depending on the treatment arm, subjects will either receive BLU-U exposure or not. Treatment arms A and B have BLU-U exposure and treatment arm C does not.
- B. Combination Arm: This treatment arm combines standard of care BLU-U exposure and daylight exposure. This treatment arm includes: Acetone preparation, ALA topical application, 15 minute incubation, 16:40 BLU-U exposure, application of sunscreen, 45 minute daylight exposure.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: BLU-U blue light phototherapy illuminator
  Aminolevulinic Acid Topical 20% Topical Solution: PDT involves the topical application of aminolevulinic acid (ALA), or one of its derivatives, as a photosensitizing agent. Subjects will receive ALA in all treatment arms (A, B, and C).
  BLU-U blue light phototherapy illuminator: Depending on the treatment arm, subjects will either receive BLU-U exposure or not. Treatment arms A and B have BLU-U exposure and treatment arm C does not.
- C. Daylight Arm: This is the experimental arm. This treatment arm includes: Acetone preparation, ALA topical application, 15 minute incubation, application of sunscreen, 1 hour daylight exposure.
  Drug intervention: Aminolevulinic acid HCl (ALA) topical solution 20% Device: none
  Aminolevulinic Acid Topical 20% Topical Solution: PDT involves the topical application of aminolevulinic acid (ALA), or one of its derivatives, as a photosensitizing agent. Subjects will receive ALA in all treatment arms (A, B, and C).
Period: Overall Study
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Started | 8 | 8 | 8
Completed | 8 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3
  >=65 years | 7 | 7 | 7 | 21
Age, Continuous [Mean (Full Range); unit: years] | 71.9 [64.4 to 85.1] | 77.7 [64.5 to 89.6] | 75.0 [60.7 to 93.9] | 75 [60 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 8 | 7 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 24
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 24
Treatment Area [Count of Participants; unit: Participants]
  Face | 5 | 6 | 6 | 17
  Scalp | 3 | 2 | 2 | 7
Actinic Keratosis Count [Mean (Standard Deviation); unit: lesion count] | 12.1 (4.2) | 11.3 (3.0) | 10.3 (3.7) | 10.8 (4.9)

OUTCOME MEASURES:

1. Primary Outcome: Change in Treatment Symptoms
Description: Primary objective is to determine whether daylight PDT changes treatment symptoms of pain, stinging/burning, and itching/pruritus. This was measured using a visual analog scale from 0-10, with higher scores indicating worse treatment symptoms, or more pain/burning/itching. Lower scores indicate less pain, burning/stinging, and itching/pruritus. Positive numbers represent increases in symptoms and negative numbers represent decreases.
Time Frame: 12 weeks
Population: 24 participants enrolled in the study who underwent treatment were analyzed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 3.9 [3.11 to 4.63] | 0.5 [-0.26 to 1.26] | 0.37 [-0.38 to 1.13]

2. Secondary Outcome: Percent Change in AK Lesion Count
Description: The number of actinic keratoses within the treatment area was counted both pre and post-treatment. Then, the mean percent change from baseline actinic keratosis lesion count was calculated for each treatment group.
Time Frame: 12 weeks
Population: 24 participants who underwent treatment were analyzed, with the data for the 1 participant in group C who was lost-to-follow up carried forward. This means that data for 8 participants in each subgroup and 24 participants overall was analyzed for this outcome.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Number analyzed (Participants) | 8 | 8 | 8
percent change | 63.9 (24.9) | 66.4 (29.5) | 61.8 (59.9)

3. Secondary Outcome: Reduction of AK Counts
Description: The number of AK lesions within the treatment area was assessed both pre and post-treatment. Then, the number of participants with various levels of AK lesion reduction (100% reduction or greater than 75% reduction) was calculated for each treatment group. This outcome measures the proportion of subjects with complete (100%) and partial (greater than or equal to 75%) reduction of baseline actinic keratosis lesion counts at 12 weeks (study end).
Time Frame: 12 weeks
Population: 24 participants who underwent treatment were analyzed, with data from the 1 participant in group C who was lost to follow up carried forward. 8 Participants were included in data analysis for each subgroup, with 24 participants included overall.
Measure: Count of Participants; unit: Participants
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Partial Clearance | 2 | 3 | 5
  Complete Clearance | 2 | 2 | 2

4. Secondary Outcome: Change in Local Skin Reaction From Pre-treatment to 12 Weeks Post-treatment
Description: To determine whether daylight PDT affords a reduction in local skin reaction to treatment. A Local Skin Response Assessment scale will be used to measure this outcome. The investigators will grade categories including Erythema, Flaking/Scaling, crusting, swelling, Pustulation (pustules), and Erosion, on a 0-4 scale (total maximum score of 24). A higher score indicates more erythema, flaking, crusting, etc. and therefore a more robust skin reaction. A score of 0 represents no erythema, flaking, crusting, etc.
Time Frame: 12 weeks
Population: 24 participants who underwent treatment were analyzed, with data from the 1 participant lost to follow up in Group C carried forward. 8 participants were analyzed for each subgroup, with 24 participants analyzed overall.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 1.0 [0.12 to 1.88] | 1.25 [0.37 to 2.13] | 1.0 [0.07 to 1.93]

5. Secondary Outcome: Peak Pain Score at Day 8 Post-treatment
Description: Pain was measured by patient report with a visual analog scale from 0-10. 0 indicates no pain and 10 indicates the maximum pain score.
Time Frame: 8 days post-treatment
Population: 24 participants who underwent treatment were analyzed, with data from the 1 participant from Group C who was lost to follow up carried forward. 8 participants from each subgroup were analyzed, with 24 participants overall. Mean peak pain on day 8 with a 95% confidence interval for each treatment group on day 8 is reported below.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
Number analyzed (Participants) | 8 | 8 | 8
score on a scale | 3.5 [2.62 to 4.38] | 5.13 [4.25 to 6.00] | 4.00 [3.07 to 4.93]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from enrollment of first participant in Decomber 2017 through completion of final participant in September 2018. Adverse events were monitored for each patient from treatment up until 84 days following treatment.
Description: Adverse events were collected at study visits by asking the participants and eliciting any relevant patient-reported adverse event information. Adverse events were defined using Common Terminology Criteria version 5.0.
Arm/Group | A. Conventional Arm | B. Combination Arm | C. Daylight Arm
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 8/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A. Conventional Arm (N=8) | B. Combination Arm (N=8) | C. Daylight Arm (N=8)
Pruritus in Treatment Area (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5) | 3 (3)
Burning/Pain in Treatment Area (Skin and subcutaneous tissue disorders) | 5 (5) | 1 (1) | 3 (3)
Scaling (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3)
Erythema in Treatment Area (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
This was a small, 24 person pilot study performed at the San Francisco Veterans Affairs Medical Center. As such, the study was not powered to detect statistically significant differences in treatment efficacies.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/93/NCT03322293/Prot_SAP_000.pdf